CLINICAL TRIAL: NCT02153645
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind, 16 Week Study to Evaluate the Efficacy and Safety of Amantadine HCl Extended Release Tablets in Parkinson's Disease Subjects With Levodopa-Induced Dyskinesias
Brief Title: Efficacy and Safety of Amantadine Hydrochloride (HCl) ER Tablets to Treat Parkinson's Disease Patients With LID.
Acronym: ALLAY-LID-I
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Adamas Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OS320-3005
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Parkinson's Disease; Levodopa Induced Dyskinesias (LID)
Keywords: Parkinson's Disease; Levodopa Induced Dyskinesias (LID); Dyskinesias; Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Dyskinesias; Parkinsonian Disorders | interventions — Amantadine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 240mg Amantadine HCl ER tablets (Experimental): Amantadine HCl ER Tablets 240mg daily for 12 weeks post two week titration phase.
  Interventions: Drug: 240mg Amantadine HCl ER tablets
- 320mg Amantadine HCl ER tablets (Experimental): Amantadine HCl ER Tablets 320mg daily for 12 weeks post a two week dose titration phase.
  Interventions: Drug: 320mg Amantadine HCl ER tablets
- Placebo tablets (Placebo Comparator): Placebo Tablets matching Amantadine HCl ER Tablets taken daily for 16 weeks.
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: 240mg Amantadine HCl ER tablets
  Other Names: Osmolex ER 240 mg Tablet
  Arms: 240mg Amantadine HCl ER tablets
Drug: Placebo tablets
  Arms: Placebo tablets
Drug: 320mg Amantadine HCl ER tablets
  Other Names: Osmolex ER 320mg Tablet
  Arms: 320mg Amantadine HCl ER tablets

SUMMARY:
This study was terminated early due to slow enrollment with 87 of 162 planned subjects enrolled. The purpose of this multi-center, randomized, double-blind, parallel-group, 16 week study is to compare the efficacy and safety of two different dose levels of Amantadine Extended Release Tablets to placebo for the treatment of levodopa induced dyskinesia in patients with Parkinson's disease.

DETAILED DESCRIPTION:
This study was terminated early due to slow enrollment with 87 of 162 planned subjects enrolled. Amantadine has been used for many years as a treatment for Parkinson's disease. It has been reported in the literature to effectively treat the motor complications of levodopa, especially dyskinesia, but it must be given 2 to 4 times a day. The purpose of this multi-center, randomized, double-blind, parallel-group, 16 week study is to compare the efficacy and safety of two different dose levels of Amantadine Extended Release Tablets to placebo for the treatment of levodopa induced dyskinesia in patients with Parkinson's disease. The dose will be given once a day in the morning so that amantadine concentrations are maintained throughout the day for treating the levodopa induced dyskinesia, but will be lower during the night, potentially reducing the negative impact of amantadine on sleep.

ELIGIBILITY:
Inclusion Criteria:

* Signed Investigational Review Board/Independent Ethics Review Committee (IRB/IEC) informed consent form.,
* Idiopathic Parkinson's disease per the United Kingdom (UK) Parkinson's Disease Society Brain Bank criteria.
* Male or female 30 to 85 years old.
* Levodopa induced, predictable peak-effect dyskinesia considered problematic and/or disabling.
* Screening serum creatinine level within normal range
* On stable doses of all oral anti-Parkinson's medication, including any levodopa preparation, for 30 days and be willing to remain on the same doses throughout the trial.
* The subject/caregiver must demonstrate the ability to complete an accurate home diary based on training and evaluation during the screening period.

Exclusion Criteria:

* Secondary parkinsonian syndrome, such as vascular, postinflammatory,drug-induced, neoplastic and post-traumatic parkinsonism or any atypical parkinsonian syndrome (e.g., Progressive Supranuclear Palsy, Multi-System Atrophy, etc.);
* Use of amantadine within 14 days before study start, or previously had an adverse event to amantadine
* Currently taking neuroleptics and atypical antipsychotic agents, acetylcholinesterase inhibitors, apomorphine, rimantadine, memantine and dextromethorphan and quinidine if used in combination for treating dyskinesia.
* History of neurosurgical intervention for treating Parkinson's s disease (i.e. pallidotomy or implanted with a deep brain stimulator).
* Any medical condition or past medical history that would increase the risk of exposure to Amantadine HCl Extended Release Tablets or interfere with safety and efficacy evaluations.
* History of cancer within 5 years of screening with following exceptions: adequately treated non-melanomatous skin cancers, localized bladder cancer, non-metastatic prostate cancer or in situ cervical cancer.
* History or current diagnosis of schizophrenia or bipolar disorder;
* Inadequately treated Major Depressive Disorder. Subjects on stable doses of selective serotonin reuptake inhibitors (SSRIs) or serotonin-norepinephrine reuptake inhibitors (SNRIs) are eligible for the study.
* Is at imminent risk of suicide or had a suicide attempt within 6 months of screening
* History or current diagnosis of Impulse Control Disorder
* Calculated plasma creatinine clearance of <60 mL/min at screening
* History of or currently has any of the following clinically significant conditions, cardiovascular, respiratory, renal, hepatic, or gastrointestinal disease
* Any clinically significant vital sign, ECG, or laboratory abnormalities:
* A positive test for HIV antibody or history of HIV; hepatitis B surface antigen unless the positive test followed a recent (<28 days) vaccination for hepatitis B; hepatitis C antibody.
* A positive urine drug test.
* Pregnant or breastfeeding at screening or has a positive pregnancy test
* If a sexually active female, is not surgically sterile or at least 2 years post-menopausal, or does not agree to utilize an effective method of contraception from the screening visit to at least 4 weeks after the completion of study treatment.
* History of alcohol or narcotic substance abuse ≤1 year before screening.
* Has dementia or another psychiatric illness that prevents provision of informed consent.
* Has a known hypersensitivity to the study treatment(s), based on known allergies to drugs of the same class including rimantadine HCl and memantine HCl.
* Has participated in other studies involving investigational drugs or surgeries within the last 30 days or investigational biologics within the last 6 months prior to screening.
* Plans to undergo major elective surgery during the course of the study.
* Received administration of Live Attenuated Influenza Vaccine (LAIV) within 2 weeks.
* Cognitive impairment, as evidenced by a score <26 on the Montreal Cognitive Assessment (MoCA) at the screening visit.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-08-18 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dentiste, MBA, Study Chair — Osmotica Pharmaceutical US LLC
Locations (51):
- United States (24):
  - Tucson, Arizona
  - Fountain Valley, California
  - Irvine, California
  - Pasadena, California
  - Reseda, California
  - Ventura, California
  - Boulder, Colorado
  - Hollywood, Florida
  - Miami, Florida
  - North Palm Beach, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Baton Rouge, Louisiana
  - Ann Arbor, Michigan
  - Summit, New Jersey
  - Brooklyn, New York
  - Manhasset, New York
  - Patchogue, New York
  - Raleigh, North Carolina
  - Columbus, Ohio
  - Round Rock, Texas
  - Orem, Utah
  - Kirkland, Washington
- Canada (2):
  - London, Ontario
  - Ottawa, Ontario
- France (12):
  - Rennes, Ille-et-Vilaine
  - Amiens
  - Bron
  - Clermont-Ferrand
  - Créteil
  - Lille
  - Marseille
  - Montauban
  - Nîmes
  - Paris
  - Poitiers
  - Toulouse
- Germany (7):
  - Haag, Bavaria
  - Erbach im Odenwald, Hesse
  - Achim, Lower Saxony
  - Bochum, North Rhine-Westphalia
  - Weissensee, State of Berlin
  - Berlin
  - Würzburg
- Spain (6):
  - Manresa, Barcelona
  - Seville, Barcelona
  - Alcorcón, Madrid
  - Castellana, Madrid
  - Barcelona
  - Pamplona

RESULTS

PARTICIPANT FLOW:
Groups:
- 240mg Amantadine Hydrochloride (HCl) ER Tablets: Amantadine HCl ER Tablets 240mg daily for 12 weeks post two week titration phase.
  Amantadine ER Tablets
- 320mg Amantadine HCl ER Tablets: Amantadine HCl ER Tablets 320mg daily for 12 weeks post a two week dose titration phase.
  Amantadine ER Tablets
- Placebo Tablets for Amantadine: Placebo Tablets matching Amantadine HCl ER Tablets taken daily for 16 weeks.
  Placebo Tablets for Amantadine ER Tablets
Period: Overall Study
Arm/Group | 240mg Amantadine Hydrochloride (HCl) ER Tablets | 320mg Amantadine HCl ER Tablets | Placebo Tablets for Amantadine
Started | 30 | 29 | 28
Completed | 17 | 19 | 18
Not Completed | 13 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- 240mg Amantadine HCl ER Tablets: Amantadine HCl ER Tablets 240mg daily for 12 weeks post two week titration phase.
  Amantadine ER Tablets
- Total: Total of all reporting groups
Arm/Group | 240mg Amantadine HCl ER Tablets | 320mg Amantadine HCl ER Tablets | Placebo Tablets for Amantadine | Total
Number analyzed (Participants) | 30 | 29 | 28 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 28 | 87
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (8.02) | 63.3 (9.17) | 66.1 (8.04) | 66.1 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 12 | 38
  Male | 14 | 19 | 16 | 49
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 0 | 1 | 2
  United States | 7 | 16 | 8 | 31
  France | 8 | 8 | 10 | 26
  Germany | 6 | 3 | 3 | 12
  Spain | 8 | 2 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Unified Dyskinesia Rating Scale
Description: The Unified Dyskinesia Rating Scale is a validated tool for assessment of dyskinesia (involuntary movements) in Parkinson's Disease patients. Rating consists of the change from baseline to Day 98 of the sum of the 26 questions comprising the questionnaire. Each question in the questionnaire is rated on a 5 point scale from 0-4 where 0 is a better outcome. Questions assess: over the past week total hours with dyskinesia and total hours without dyskinesia; problems with speech, chewing and swallowing, eating, dressing, hygiene, handwriting, hobbies, balance, socializing, emotions, spasm or cramps, pain without dystonia (spasm or cramps) and pain from dystonia, the degree of impairment for each of 7 body parts, and the degree of disability in communication, drinking from a cup, dressing and ambulation. The minimum score is 0 (better) and the maximum score is 130 (worse).
Time Frame: From baseline to Day 98
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 240 mg Amantadine HCl ER Tablets: Amantadine HCl ER Tablets 240 mg daily for 12 weeks post two week titration phase.
  Amantadine ER Tablets
- 320 mg Amantadine HCl ER Tablets: Amantadine HCl ER Tablets 320 mg daily for 12 weeks post two week titration phase.
  Amantadine ER Tablets
- Placebo Amantadine HCl ER Tablets: Amantadine HCl ER Placebo Tablets daily for 12 weeks post two week titration phase.
  Amantadine ER Tablets
Arm/Group | 240 mg Amantadine HCl ER Tablets | 320 mg Amantadine HCl ER Tablets | Placebo Amantadine HCl ER Tablets
Number analyzed (Participants) | 30 | 29 | 28
score on a scale
  Visit 2 (Baseline) | 46.2 (13.19) | 39.2 (11.91) | 38.7 (11.23)
  Visit 7 (Day 98)/Stable Dose LOCF [1] | 27.5 (19.13) | 26.4 (13.17) | 28.7 (13.70)
  Change from Baseline (SD) | -18.8 (16.38) | -13.3 (13.73) | -9.6 (14.87)
Statistical Analysis 1: Comparison: 240 mg Amantadine HCl ER Tablets vs 320 mg Amantadine HCl ER Tablets vs Placebo Amantadine HCl ER Tablets; Test type: Superiority or Other; p = 0.179, ANCOVA; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-13.9 to 2.6], Standard Error of Mean 2.90
Statistical Analysis 2: Comparison: 320 mg Amantadine HCl ER Tablets; Test type: Superiority; p = 0.458, ANCOVA; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-11.2 to 5.1], Standard Error of Mean 2.95

2. Secondary Outcome: Mobility State Self-Assessment - Subject Diary Cards
Description: Change from baseline in the number of awake hours without troublesome dyskinesia (involuntary movements). Every half hour the subject will indicate in the diary if the medication has ("ON") or has not ("OFF") produced benefits in terms of mobility, slowness and rigidity. Valid diaries of the 3 consecutive days prior to each visit will be averaged with respect to the number of awake hours without troublesome dyskinesia. The change from baseline in the number of waking hours that subjects report being "ON" without troublesome dyskinesias will be analyzed at analysis visits Day 14 and Day 98 of treatment. Higher scores mean a better outcome and the maximum value is 24 hours.
Time Frame: Day 14 and Day 98 of treatment
Population: The number analyzed was the number of subjects with values at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 240 mg Amantadine HCl ER Tablets | 320 mg Amantadine HCl ER Tablets | Placebo Amantadine HCl ER Tablets
Number analyzed (Participants) | 30 | 29 | 28
score on a scale
  Visit 2 (Baseline): number analyzed (Participants) | 26 | 25 | 19
  Visit 2 (Baseline) | 3.5 (2.02) | 3.3 (2.63) | 4.3 (2.59)
  Visit 7 (Day 98)/Stable Dose LOCF [1]: number analyzed (Participants) | 30 | 27 | 25
  Visit 7 (Day 98)/Stable Dose LOCF [1] | 4.1 (2.48) | 2.8 (2.24) | 3.8 (2.36)
  Change from Baseline (SD): number analyzed (Participants) | 30 | 27 | 25
  Change from Baseline (SD) | 0.8 (2.92) | -0.5 (2.18) | 0.1 (2.78)

ADVERSE EVENTS:
Time Frame: Three months
Arm/Group | 240mg Amantadine HCl ER Tablets | 320mg Amantadine HCl ER Tablets | Placebo Tablets for Amantadine
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/30 | 1/29 | 2/28
Other Adverse Events (participants affected / at risk) | 20/30 | 24/29 | 15/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 240mg Amantadine HCl ER Tablets (N=30) | 320mg Amantadine HCl ER Tablets (N=29) | Placebo Tablets for Amantadine (N=28)
syncope (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
traumatic haemothroax (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
megacolon multi-organ failure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
arthralgia osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
impulse-control disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 240mg Amantadine HCl ER Tablets (N=30) | 320mg Amantadine HCl ER Tablets (N=29) | Placebo Tablets for Amantadine (N=28)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 4 (4) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure orthostatic (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine ketone body present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Akinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndorme (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Dyskinesia (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Freezing phenomenon (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
On and off phenomenon (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 4 (4) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersexuality (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Illusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Impulse-control disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep attacks (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatism (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Gambling (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall allow SPONSOR 60 days to review any manuscript and 30 days to review any poster presentation, abstract or any other written or oral material which discloses the Study Results. SPONSOR may request in writing an additional 60 days for review.

SPONSOR may remove all Confidential Information from any publications or presentations, or if deemed not sufficient to protect its Intellectual Property Rights, then SPONSOR may embargo the publication or presentation.